CLINICAL TRIAL: NCT06053801
Title: A Real-world, Prospective, Multicenter Study of Safety and Effectiveness of Xolair® (Omalizumab) in the Treatment of Chronic Spontaneous Urticaria (CSU) in Chinese Adolescents Inadequately Controlled With H1 Antihistamines
Brief Title: A Real-world Study to Assess Safety and Effectiveness of Xolair® in Pediatric Chronic Spontaneous Urticaria in China
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025ECN01
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic Spontaneous Urticaria; CSU; PASS; Omalizumab; Chinese
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xolair: Chinese adolescents with Chronic Spontaneous Urticaria (CSU) inadequately controlled with H1 antihistamines
  Interventions: Other: Xolair

INTERVENTIONS:
Other: Xolair — Prospective observational cohort study. There is no treatment allocation. Patients administered Xolair by prescription will be enrolled.
  Other Names: Omalizumab

SUMMARY:
This non-interventional, multi-center, prospective post-approval study aims to provide safety and effectiveness data of Xolair® in Chinese adolescents with Chronic Spontaneous Urticaria who remain symptomatic despite H1 antihistamine treatment. The study period is 16 weeks which contains a 12-week treatment period and 4-week safety follow-up.

DETAILED DESCRIPTION:
The study period is 16 weeks which contains a 12-week treatment effect evaluation period and 4-week safety follow up. The primary objective is to evaluate the safety of Xolair® in a real-world setting in Chinese adolescent patients with Chronic Spontaneous Urticaria who remain symptomatic despite H1 antihistamine treatment over a 16-week study period. The secondary objectives are to evaluate the effectiveness (measured by ISS7, UAS7, UCT) of Xolair® and the quality of life (measured by CDLQI) of Chinese adolescent patients over a 12-week treatment period. Data will be collected in conjunction with routine care visits at the site, at Week 4, 8, 12 (recommended scheduled visits). Routine clinical assessments will be conducted, and safety information will be collected. Safety information includes AE/SAE collection, including but not limited to lab tests, vital signs, weight, physical examination etc. No extra study visits, examinations, laboratory tests or procedures other than activities performed in clinical practice will be mandated.

ELIGIBILITY:
Inclusion Criteria:

The patient should meet all of the following criteria:

1. Diagnosed with CSU refractory to H1-AH at approved doses as defined by all of the following:

   * The presence of itch and hives for ≥ 6 consecutive weeks at any time prior to enrollment despite current use of second-generation H1-AH (at locally approved doses)
   * UAS7 score (range 0-42) ≥ 16 and ISS7 (range 0-21) ≥ 8 as captured in the UPDD during the 7 days prior to treatment initiation with Xolair®
2. Willing and able to complete a daily symptom Diary (UPDD) for the duration of the study, and having no more than 3 missing diary entries in the screening period.
3. Planned to receive Xolair® treatment according to the approved label in China at the time of screening.

Exclusion Criteria:

The patient should not meet any of the following criteria:

1. Use of other investigational drugs for CSU treatment within 5 half-lives, or within 30 days (for small molecules) prior to screening or until the expected pharmacodynamic effect has returned to baseline (for biologics), whichever is longer.
2. History of hypersensitivity to any of the anti-IgE drugs or their excipients or to drugs of similar classes (i.e. to murine, chimeric, or human antibodies).
3. Any other skin disease associated with chronic itching that might influence, in the investigators opinion, the study evaluations and results. (e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.)

Other protocol-defined inclusion/exclusion criteria may apply at the end.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Chinese pediatric patients aged between 12 to less than 18 years and diagnosed with Chronic Spontaneous Urticaria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
AE/AESI/SAE type and frequency | 16 weeks
  The type and frequency of adverse event (AE), adverse events of special interest (AESI) and serious adverse event (SAE) will be used as variables to evaluate the primary objective. AESI terms include Anaphylaxis, Churg Strauss Syndrome, Arterial Thromboembolic Events and Malignant neoplasms.

SECONDARY OUTCOMES:
ISS7 (weekly Itch Severity Score) | 12 weeks
  A weekly itch score is derived by adding up the average daily ISS of the 7 days preceding the visit. ISS is ranged on a scale of 0 (none) to 3 (intense/severe), therefore, the possible range of the ISS7 is 0 to 21 where higher scores indicate more intense itch.
UAS7 (Weekly Urticaria Severity Score) | 12 weeks
  The number of hives and intensity of itch score will be recorded by the patient in Urticaria Patient Daily Diary (UPDD), on a scale of 0 (none) to 3 (intense/severe). The Urticaria Severity Score (UAS) is a composite score of the number of wheals (hives) (Hives Severity Scores, HSS); and the severity of the itch (Itch Severity Scores, ISS). A weekly hives score (HSS7) is derived by adding up the average daily HSS of the 7 days preceding the visit. The possible range of the HSS7 is therefore 0 to 21. A weekly itch score (ISS7) is derived by adding up the average daily ISS of the 7 days preceding the visit. The possible range of the ISS7 is therefore 0 to 21. The UAS7 is the sum of the HSS7 score and the ISS7 score. The possible range of the weekly UAS7 score is 0 to 42 (highest activity).
Urticaria Control Test (UCT) score | 12 weeks
  Frequency and percentage will be provided for patients who achieved well-controlled CSU (defined as a UCT score ≥12) at Week 12.
  The UCT is a 4-item Patient Reported Outcome measure developed to assess disease control in patients with Chronic Urticaria specifically Chronic Spontaneous Urticaria and Chronic Inducible Urticaria. It has a 7 days recall period and patients respond with how much they were bothered by their urticaria symptoms, what is the impact on QoL, how often the treatment did not control their urticaria and their overall perception of disease control. Each question can be scored on a scale from 0 to 4 and the overall score ranges from 0 (no control) to 16 (maximum control). The cut-off value for disease control was established at 12. Patients with a score above 12 are considered controlled. A minimally important difference of 3 points was validated as reflective of a clinically relevant change of control
Proportion of patients achieving Children's Dermatology Life Quality Index (CDLQI) 0 or 1 over time | 12 weeks
  The Children's Dermatology Life Quality Index is a 10-item general dermatology disability index designed to assess health-related quality of life in pediatric subjects aged 4 to 16 years. It is self-explanatory and may be completed by the child with assistance from parents or caregivers as necessary. The 10 questions cover six areas of daily activities including symptoms and feelings, leisure, school or holidays, personal relationships, sleep and treatment. The questions are based on the preceding week to permit accurate recall. Each question is answered on a 4-point Likert scale scored from 0 to 3. These are added to give a minimum score of 0 and maximum score of 30. A higher CDLQI score indicates a greater degree of QoL impairment. The CDLQI questionnaire will be completed by all patients independent of age, to ensure consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- China (9):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18413